CLINICAL TRIAL: NCT00608205
Title: A Phase III Randomized Trial Comparing Single Agent Cisplatin With the Combination of 5-Fluorouracil and Cisplatin, Concurrent With Radiation Therapy in Stage III and IV Squamous Cell Head and Neck Cancer
Brief Title: Radiation Therapy Cisplatin With or Without Fluorouracil Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3307; NCI-2010-01197 (Other: NCI/CTRP)
Record Dates: First submitted 2008-01-30; First posted 2008-02-06 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Radiation with concurrent Cisplatin (Active Comparator): Patients undergo full-dose radiotherapy once or twice daily 5 days a week for up to 7 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
  Interventions: Drug: cisplatin; Radiation: radiation therapy
- Arm B: Radiation with concurrent 5-FU and Cisplatin (Experimental): Patients undergo radiotherapy as in arm I and receive fluorouracil IV and cisplatin IV continuously on days 1-4 and 22-25 of radiotherapy.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CDDP
Drug: fluorouracil — Given IV
  Arms: Arm B: Radiation with concurrent 5-FU and Cisplatin
Radiation: radiation therapy — Patients undergo full-dose radiotherapy once or twice daily 5 days a week for up to 7 weeks
  Other Names: radiation

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with cisplatin and fluorouracil may kill more tumor cells. It is not yet known whether radiation therapy and cisplatin are more effective with or without fluorouracil in treating patients with head and neck cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy and cisplatin to compare how well they work with or without fluorouracil in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the relapse-free survival of patients treated with radiotherapy and cisplatin with vs without fluorouracil.
* To compare the overall survival, local control without surgery, and patterns of failure in patients treated with these regimens.
* To compare the acute and long-term toxicity of these regimens in these patients.
* To compare the quality of life of patients treated with these regimens.
* To prospectively collect biopsy material, mucosal scrapings, and serum in an effort to generate hypotheses for future correlative studies.

OUTLINE: This is a multicenter study. Patients are stratified according to radiotherapy schedule (once daily vs twice daily) and radiotherapy planning (2D vs 3D vs intensity-modulated radiotherapy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo full-dose radiotherapy once or twice daily 5 days a week for up to 7 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
* Arm II: Patients undergo radiotherapy as in arm I and receive fluorouracil IV and cisplatin IV continuously on days 1-4 and 22-25 of radiotherapy.

Patients with biopsy-verified residual disease at the primary site or local recurrence after achieving a complete response to chemoradiotherapy may undergo salvage surgery 12 weeks after the completion of chemoradiotherapy.

Patients complete questionnaires periodically to assess late toxicity and quality of life.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx

  * No histologic diagnosis other than squamous cell carcinoma
  * A primary site must be identified
* Must have locoregionally confined stage III (excluding T1-2, N1) or stage IV disease

  * No evidence of nodal disease below the clavicles or distant hematogenous metastases (M0)
  * No stage IVC disease (stage IVB disease allowed)
* Deemed appropriate for definitive non-operative management with curative intent

  * Resectable disease is not required
* No primary cancer of the nasopharynx, paranasal sinus, or salivary gland

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 3,500/mm³
* Platelet count > 100,000/mm³
* Serum creatinine < 2.0 mg/dL
* Alkaline phosphatase < 2 times normal
* AST < 2 times normal
* Bilirubin ≤ 2.0 mg/dL
* Serum calcium normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No unstable or uncontrolled angina
* No clinically apparent jaundice
* No active infection
* No history of any other malignancy (except squamous cell or basal cell skin cancer or cervical carcinoma in situ), unless the patient has been continuously disease-free for at least 5 years
* Not a poor compliance risk
* Able to withstand the rigors of intensive treatment
* Available for and compliant with adequate long-term follow-up

PRIOR CONCURRENT THERAPY:

* No prior definitive surgery or radiotherapy for this malignancy
* No prior chemotherapy, immunotherapy, or epidermal growth factor receptor inhibitors for any disease Patients who have had previous definitive surgery, or radiation therapy for this malignancy, and patients who have had any previous chemotherapy, immunotherapy, or EGF receptor inhibition for any disease are ineligible.

Exclusion Criteria Patients with primary cancers of the nasopharynx, paranasal sinus or salivary gland are ineligible.

Patients with unstable or uncontrolled angina, clinically apparent jaundice, or active infection are ineligible.

Patients with a history of any other malignancy (except squamous or basal cell skin cancer or cervical carcinoma in-situ) are ineligible, unless the patient has been continuously disease-free for at least 5 years.

Patients with any histologic diagnosis other than squamous cell carcinoma are ineligible.

Patients who might be a poor-compliance risk are ineligible.

Pregnant or breastfeeding women are ineligible. Women/men of reproductive potential must be willing to practice acceptable methods of birth control to prevent pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-01; Primary Completion 2012-09 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Panayiotis Savvides, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from Cleveland, Ohio medical clinics from December 2007 to August 2012.
Period: Overall Study
Arm/Group | Arm A: Radiation With Concurrent Cisplatin | Arm B: Radiation With Concurrent 5-FU and Cisplatin
Started | 35 | 34
Completed | 32 | 31
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 2
Not completed — Patient non-compliant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Radiation With Concurrent Cisplatin | Arm B: Radiation With Concurrent 5-FU and Cisplatin | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Customized [Number; unit: participants]
  40-49 years | 6 | 10 | 16
  50-59 years | 11 | 16 | 27
  60-69 years | 17 | 6 | 23
  70-79 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 35 | 33 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Number of patients that are alive without recurrence when recurrence is defined by any subject with new evidence of cancer after achieving a complete response. Complete response is defined by the complete disappearance of all clinically and radiologically detectable tumor..
Time Frame: at 2 yrs from start of study
Population: intention to treat (ITT)
Measure: Number; unit: participants
Groups:
- Arm A: Patients undergo full-dose radiotherapy once or twice daily 5 days a week for up to 7 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
- Arm B: Patients undergo radiotherapy as in arm I and receive fluorouracil IV and cisplatin IV continuously on days 1-4 and 22-25 of radiotherapy.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 34
participants | 30 | 28

2. Secondary Outcome: Patterns of Failure
Description: Patients with any new evidence of cancer after achieving a complete response are considered to have recurrent disease. Biopsy verification will be obtained if at all possible and salvage surgery is recommended if possible. Disease recurrence will be characterized as either local, regional(nodal) or distant recurrence. Patients may have more than one kind of recurrence.
Time Frame: 2 years from start of study
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 34
participants
  Local recurrence | 1 | 1
  Regional (nodal) recurrence | 1 | 0
  Distant recurrence | 4 | 4

3. Secondary Outcome: Overall Survival
Description: Number of patients still alive from 2 years from start of study
Time Frame: 2 yrs from start of study
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 34
participants | 34 | 29

4. Secondary Outcome: Number of Patients With a Clinical Response-complete Disappearance of Detectable Tumor
Description: Twelve weeks after completing chemoradiotherapy, a formal evaluation for response will be made, to include a careful evaluation by the head and neck surgeon, medical and radiation oncologists, and, as appropriate, a radiologic and an endoscopic examination. Patients will be considered to have achieved either a clinical complete response (i.e. complete disappearance of all clinically and radiologically detectable tumor) or to have clinical persistent disease.
Time Frame: at 12 weeks after completing chemoradiotherapy
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 34
participants | 35 | 28

5. Secondary Outcome: Number of Patients With a Pathological(Final)Complete Response
Description: A Pathological, or final response will be assigned to subjects after any salvage surgery is performed for clinical persistent disease, and after planned neck dissection in those achieving a clinical complete response. If no surgery is performed after chemoradiotherapy, the clinical and pathological (final) response will be the same. Patient will be coded as having either a pathologic complete response, or as having pathologic persistent disease. A pathologic complete response will be defined as the total disappearance of all clinically and radiologically detectable tumor.
Time Frame: at 12 weeks after completing chemoradiotherapy and surgery
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 34
participants | 35 | 31

6. Secondary Outcome: Disease Recurrence
Description: Number of patients with any new evidence of cancer after achieving a complete response (at 12 weeks after completing chemoradiotherapy) are considered to have recurrent disease.
Time Frame: 2 years after start of study
Population: Patients that had a complete response after 12 weeks of therapy
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 35 | 31
participants | 5 | 2

7. Secondary Outcome: Number of Patients That Required a Feeding Tube
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 29 | 26
participants | 0 | 3

8. Secondary Outcome: Number of Patients That Required a Feeding Tube
Time Frame: 8 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 24
participants | 0 | 0

9. Secondary Outcome: Number of Patients That Required a Feeding Tube
Time Frame: 12 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 23
participants | 0 | 0

10. Secondary Outcome: Number of Patients That Required a Feeding Tube
Time Frame: 24 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 21 | 17
participants | 0 | 0

11. Secondary Outcome: Nausea Level
Description: Quality of life questionnaire asking "I have nausea".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4).
  N (number of patients analyzed) is based on number of patients who completed the question.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 26
units on a scale | 0.07 (0.26) | 0.12 (0.33)

12. Secondary Outcome: Nausea Level
Description: Quality of life questionnaire asking "I have nausea".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 8 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 0.15 (0.46) | 0.09 (0.29)

13. Secondary Outcome: Nausea Level
Description: as for outcome 12
Time Frame: 12 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 23
units on a scale | 0.14 (0.45) | 0.04 (0.21)

14. Secondary Outcome: Nausea Level
Description: Quality of life questionnaire asking "I have nausea".
Time Frame: 24 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Radiation With Concurrent Cisplatin: Patients undergo full-dose radiotherapy once or twice daily 5 days a week for up to 7 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
- Radiation With Concurrent 5-FU and Cisplatin: Patients undergo radiotherapy as in arm I and receive fluorouracil IV and cisplatin IV continuously on days 1-4 and 22-25 of radiotherapy.
Arm/Group | Radiation With Concurrent Cisplatin | Radiation With Concurrent 5-FU and Cisplatin
Number analyzed (Participants) | 21 | 16
units on a scale | 0.10 (0.3) | 0 (0)

15. Secondary Outcome: Dry Mouth
Description: Quality of life questionnaire asking "My mouth is dry".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 25
units on a scale | 3.33 (0.83) | 3.08 (1.15)

16. Secondary Outcome: Dry Mouth
Description: as for outcome 15
Time Frame: 8 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 2.67 (1.07) | 3.09 (0.85)

17. Secondary Outcome: Dry Mouth
Description: as for outcome 15
Time Frame: 12 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 22
units on a scale | 2.70 (1.03) | 3.09 (0.92)

18. Secondary Outcome: Dry Mouth
Description: as for outcome 15
Time Frame: 24 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 20 | 16
units on a scale | 2.60 (1.10) | 2.94 (1.29)

19. Secondary Outcome: Pain
Description: Quality of life questionnaire asking "I have pain in my mouth, throat or neck".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 29 | 26
units on a scale | 1.24 (1.06) | 1.42 (0.95)

20. Secondary Outcome: Pain
Description: as for outcome 19
Time Frame: 8 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 26 | 23
units on a scale | 0.65 (0.80) | 0.74 (0.81)

21. Secondary Outcome: Pain
Description: as for outcome 19
Time Frame: 12 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 23
units on a scale | 0.57 (0.74) | 0.57 (0.79)

22. Secondary Outcome: Pain
Description: as for outcome 19
Time Frame: 24 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 20 | 16
units on a scale | 0.60 (0.75) | 0.75 (1.00)

23. Secondary Outcome: Quality of Life
Description: Quality of life questionnaire asking "I am content with the quality of my life right now".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 25
units on a scale | 1.37 (1.08) | 1.68 (1.14)

24. Secondary Outcome: Quality of Life
Description: as for outcome 23
Time Frame: 8 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 0.85 (1.13) | 1.13 (1.18)

25. Secondary Outcome: Quality of Life
Description: as for outcome 23
Time Frame: 12 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 22
units on a scale | 0.67 (1.00) | 0.95 (0.84)

26. Secondary Outcome: Quality of Life
Description: as for outcome 23
Time Frame: 24 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 21 | 16
units on a scale | 0.62 (0.86) | 0.88 (0.81)

27. Secondary Outcome: Eating
Description: Quality of life questionnaire asking "I am able to eat the foods i like".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 25
units on a scale | 2.33 (1.07) | 2.28 (1.02)

28. Secondary Outcome: Eating
Description: as for outcome 27
Time Frame: 8 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 1.93 (1.17) | 1.78 (0.95)

29. Secondary Outcome: Eating
Description: as for outcome 27
Time Frame: 12 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 21
units on a scale | 1.56 (1.25) | 1.24 (1.09)

30. Secondary Outcome: Eating
Description: as for outcome 27
Time Frame: 24 months from start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 21 | 16
units on a scale | 1.52 (1.17) | 1.13 (1.09)

31. Secondary Outcome: Swallowing
Description: Quality of life questionnaire asking "I can swallow naturally and easily".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 29 | 26
units on a scale | 1.93 (1.07) | 2.31 (0.97)

32. Secondary Outcome: Swallowing
Description: as for outcome 31
Time Frame: 8 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 26 | 23
units on a scale | 1.31 (1.12) | 1.83 (1.03)

33. Secondary Outcome: Swallowing
Description: as for outcome 31
Time Frame: 12 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 28 | 23
units on a scale | 1.61 (1.13) | 1.52 (1.16)

34. Secondary Outcome: Swallowing
Description: as for outcome 31
Time Frame: 24 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 20 | 16
units on a scale | 1.45 (1.00) | 1.63 (1.20)

35. Secondary Outcome: Alcohol Consumption
Description: Quality of life questionnaire asking "I drink alcohol (e.g. beer, wine)".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 29 | 26
units on a scale | 3.28 (0.65) | 3.27 (0.87)

36. Secondary Outcome: Alcohol Consumption
Description: as for outcome 35
Time Frame: 8 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 25 | 23
units on a scale | 2.96 (0.89) | 3.00 (0.85)

37. Secondary Outcome: Alcohol Consumption
Description: as for outcome 35
Time Frame: 12 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 2.85 (0.72) | 2.91 (0.73)

38. Secondary Outcome: Alcohol Consumption
Description: as for outcome 35
Time Frame: 24 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 20 | 16
units on a scale | 2.85 (0.88) | 2.81 (0.66)

39. Secondary Outcome: Solid Foods
Description: Quality of life questionnaire asking "I can eat solid foods".
  The Categories were assigned a number. The categories were: Not at all (0), A little bit (1), Somewhat (2), Quite a bit (3), Very much (4). The mean was determined from each statement.
Time Frame: 12 weeks (after treatment)
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 29 | 26
units on a scale | 1.41 (1.35) | 1.73 (1.15)

40. Secondary Outcome: Solid Foods
Description: as for outcome 39
Time Frame: 8 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 26 | 23
units on a scale | 0.96 (1.15) | 1.13 (1.06)

41. Secondary Outcome: Solid Foods
Description: as for outcome 39
Time Frame: 12 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 27 | 23
units on a scale | 0.78 (0.97) | 0.70 (0.93)

42. Secondary Outcome: Solid Foods
Description: as for outcome 39
Time Frame: 24 months after start of treatment
Population: Patients still alive from Cleveland Clinic only. University Hospital patients were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 20 | 16
units on a scale | 0.85 (0.93) | 0.56 (0.89)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 2 year period from study start.
Arm/Group | Arm A: Radiation With Concurrent Cisplatin | Arm B: Radiation With Concurrent 5-FU and Cisplatin
Serious Adverse Events (participants affected / at risk) | 7/35 | 14/34
Other Adverse Events (participants affected / at risk) | 35/35 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Radiation With Concurrent Cisplatin (N=35) | Arm B: Radiation With Concurrent 5-FU and Cisplatin (N=34)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac (Cardiac disorders) | 0 | 2
Cranial Neuropathy/ Hearing and Balance (Nervous system disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 2 | 9
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Investigations) | 0 | 1
Malnutrition (Gastrointestinal disorders) | 1 | 2
Mucositis/Dysphagia (Gastrointestinal disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pain-not otherwise specified (NOS) (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Radiation With Concurrent Cisplatin (N=35) | Arm B: Radiation With Concurrent 5-FU and Cisplatin (N=34)
Cranial Neuropathy/ Hearing and Balance (Nervous system disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 33 | 34
Hypothyroidism (Endocrine disorders) | 14 | 16
Increased Creatinine (Investigations) | 9 | 1
Mucositis (Gastrointestinal disorders) | 34 | 33
Mucositis/Dysphagia (Gastrointestinal disorders) | 34 | 34
Nausea/Vomiting (Gastrointestinal disorders) | 27 | 23
Neutropenia (Blood and lymphatic system disorders) | 12 | 21
Skin Toxicity from Radiation (Injury, poisoning and procedural complications) | 33 | 30
Stomatitis (Gastrointestinal disorders) | 13 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes